CLINICAL TRIAL: NCT06447454
Title: Chemoradiotherapy Combined With Slulimumab in the Treatment of First-line Intrahepatic Cholangiocarcinoma: Efficacy and Safety Evaluation of a Phase II Clinical Study
Brief Title: Combining Chemoradiotherapy With Sintilimab in First-Line ICC
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: zs-ICC-RT+GC+HLX10
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: ICC
MeSH Terms: interventions — Radiotherapy; Gemcitabine; Cisplatin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- GC (gemcitabine + cisplatin) + radiotherapy + slulimumab Group: First-line treatment for patients with intrahepatic bile duct carcinoma involves the administration of GC (gemcitabine plus cisplatin) along with radiotherapy and sintilimab.
  Interventions: Radiation: radiotherapy; Drug: gemcitabine + cisplatin; Drug: slulimumab

INTERVENTIONS:
Radiation: radiotherapy — radiotherapy
  Other Names: RT
Drug: gemcitabine + cisplatin — Gemcitabine 1000mg/m² intravenous infusion over 30 minutes, cisplatin 25mg/m² intravenous infusion, on day 1 and day 8, every 3 weeks.
  Other Names: GC
Drug: slulimumab — Slulimumab, 4.5mg/kg intravenous infusion, Q3W
  Other Names: HLX10

SUMMARY:
To evaluate the effectiveness and safety of GC (gemcitabine + cisplatin) and radiotherapy combined with slulimumab in the treatment of first-line intrahepatic cholangiocarcinoma patients

ELIGIBILITY:
Inclusion Criteria:

1. Cholangiocarcinoma confirmed by histology/cytology.
2. The included patients were patients with first-line intrahepatic cholangiocarcinoma treated with GC (gemcitabine + cisplatin) and radiotherapy combined with slulimumab. All lesions are required to be eligible for RT treatment, and at least one of them is evaluable.
3. Liver function Child-Pugh class A, other laboratory tests:

   Neutrophils ≥1.5×109/L； Platelets ≥75×109/L；Hemoglobin ≥90g/L (no blood transfusion record within 2 weeks or no dependence on erythropoietin (EPO))；Serum creatinine ≤1.5 times ULN or calculated creatinine clearance ≥ 60 ml/min (Cockcroft-Gault formula)；AST ≤2.5×ULN, ALT ≤2.5×ULN; if intrahepatic lesions are present, ALT and AST ≤5×ULN；TSH, FT3, FT4 within ± 10% of normal values；Coagulation function: international normalized ratio (INR) ≤ 2 times ULN, and activated partial thromboplastin time (APTT) ≤ 1.5 times ULN
4. ECOG score 0-1 points.
5. Expected survival time > 3 months.
6. No history of radiation therapy.
7. Age ≥18 years old and ≤75 years old.
8. Sign the informed consent form and be able to comply with the visits and related procedures stipulated in the plan.
9. Female subjects of childbearing age or male subjects whose sexual partners are women of childbearing age must take effective contraceptive measures during the entire treatment period and for 6 months after the treatment period.

Exclusion Criteria:

1. Histology includes components such as hepatocellular carcinoma, fibrolamellar hepatocellular carcinoma, and sarcomatoid hepatocellular carcinoma.
2. Have a history of hepatic encephalopathy or liver transplantation.
3. Pleural effusion, ascites, and pericardial effusion with clinical symptoms or needing drainage, only imaging shows a small amount of pleural effusion, ascites, and pericardial effusion and are asymptomatic and can be selected.
4. People with acute or chronic active hepatitis B or hepatitis C infection, hepatitis B virus (HBV) DNA>2000IU/ml or 104 copies/ml; hepatitis C virus (HCV) RNA>103 copies/ml; hepatitis B Surface antigen (HbsAg) and anti-HCV antibodies were positive at the same time.
5. Symptomatic central nervous system metastasis. Patients with asymptomatic brain metastases or stable symptoms after treatment of brain metastases can participate in this study as long as they meet all the following criteria: measurable lesions outside the central nervous system; no midbrain, pons, cerebellum, meninges, Bulbar or spinal cord metastases; maintain clinical stability for at least 4 weeks; discontinue glucocorticoid therapy two weeks before the first dose of study drug.
6. History of gastrointestinal perforation and/or fistula, intestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), inflammatory bowel disease, or extensive intestinal resection (partial colectomy or extensive small bowel resection) within the past 6 months , complicated by chronic diarrhea), Crohn's disease, ulcerative colitis, or chronic diarrhea.
7. History of interstitial pneumonia, drug-induced pneumonia, idiopathic pneumonia or active pneumonia. Radiation pneumonitis within the radiation treatment area is permitted.
8. Active tuberculosis (TB), currently receiving anti-tuberculosis treatment or those who have received anti-tuberculosis treatment within 1 year before the first dose.
9. People infected with human immunodeficiency virus (HIV) (HIV 1/2 antibody positive).
10. Severe infection in active stage or with poor clinical control. Severe infection within 4 weeks before first dose, including but not limited to hospitalization due to complications of infection, bacteremia, or severe pneumonia.
11. Active autoimmune diseases that require systemic treatment or a history of the disease within the past 2 years (vitiligo, psoriasis, alopecia or Grave's disease that does not require systemic treatment within the past 2 years, only thyroid hormone is required Patients with hypothyroidism requiring replacement therapy and patients with type I diabetes requiring only insulin replacement therapy are eligible). Known history of primary immunodeficiency. Patients who are only positive for autoimmune antibodies need to confirm whether there is an autoimmune disease according to the researcher's judgment.
12. Use of immunosuppressive drugs within the past 4 weeks, excluding topical glucocorticoids by nasal spray, inhalation or other routes or systemic glucocorticoids at physiological doses (i.e. not exceeding 10 mg/day of prednisone or other (other glucocorticoids at effective doses), and the temporary use of glucocorticoids for the treatment of dyspnea symptoms in diseases such as asthma and chronic obstructive pulmonary disease is allowed.
13. Have received live attenuated vaccines within the past 4 weeks or plan to during the study period.
14. Have received systemic immunostimulant treatment within the past 4 weeks.
15. Received major surgical surgery (craniotomy, thoracotomy or laparotomy) or unhealed wounds, ulcers or fractures within the past 4 weeks.
16. Uncontrolled metabolic disorders or other non-malignant tumor organs or systemic diseases or secondary reactions to cancer, which may lead to higher medical risks and/or uncertainty in survival evaluation.
17. Other acute or chronic diseases, psychiatric disorders, or abnormal laboratory test values that may increase the risks associated with study participation or administration of study drugs, or interfere with the interpretation of study results, and which, at the discretion of the investigator, may cause the patient to were listed as ineligible to participate in this study.
18. Other malignant tumors diagnosed within 5 years before the first dose, excluding radically cured cutaneous basal cell carcinoma, cutaneous squamous cell carcinoma and/or radically resected carcinoma in situ. If other malignant tumors or liver cancer are diagnosed more than 5 years before administration, pathological or cytological diagnosis of recurrent and metastatic lesions is required.
19. Pregnant or breastfeeding female patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: First-line patients with intrahepatic cholangiocarcinoma
Sampling Method: Probability Sample
Enrollment: 19 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival(PFS) | 2 years
  The time from the date of first treatment to disease progression or death, whichever occurs first.

SECONDARY OUTCOMES:
Time-To-Progression | 2 years
  The time from the date of first treatment to any recorded imaging tumor progression.
Objective Response Rate | 2 years
  The use of RECIST version 1.1 standards to evaluate the objective efficacy of tumors, including cases of CR and PR.
Disease Control Rate | 2 years
  The percentage of CR, PR and SD (≥4 weeks) cases among patients whose efficacy can be evaluated.
Incidence of Adverse events | 2 years
  AEs and SAEs, drug-related AEs and SAEs.

CONTACTS AND LOCATIONS:
Overall Officials: Shisuo Du, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
The IPD will not be shared with other researchers in order to protect patients' privacy.